CLINICAL TRIAL: NCT03523442
Title: A Phase 1 Study of Androgen Receptor (AR) Antagonist Apalutamide in Chinese Subjects With Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Study of Androgen Receptor (AR) Antagonist Apalutamide in Chinese Participants With Metastatic Castration-Resistant Prostate Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR107444; 56021927PCR1013 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2018-05-02; First posted 2018-05-14 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Apalutamide (Experimental): Participants will receive a single oral dose of apalutamide 240 milligram (mg) during pharmacokinetics (PK) Week Day 1 and will be monitored for one week (that is; PK Week) to assess PK and safety of drug. Subsequently, participants will further receive daily treatment of apalutamide from Cycle 1 Day 1 onwards until disease progression, withdrawal of consent, lost to follow-up, or the occurrence of unacceptable toxicity. Each treatment cycle consists of 28 days. After final analysis (FA), participants who are receiving apalutamide in the open-label treatment phase may continue receiving single oral dose apalutamide 240 mg once daily in a long-term extension (LTE) phase if they continue to derive benefit from treatment (based on investigator assessment).
  Interventions: Drug: Apalutamide

INTERVENTIONS:
Drug: Apalutamide — The participants will receive apalutamide 240 mg once daily orally.
  Other Names: JNJ-56021927

SUMMARY:
The purpose of this study is to evaluate pharmacokinetics (PK) following a single dose and multiple dose treatment and the safety of apalutamide in Chinese participants with metastatic castration resistant prostate cancer (mCRPC) at dose of 240 milligram (mg).

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to (<=) 2
* Histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features
* Metastatic disease as documented by bone scan or metastatic lesions by computed tomography or magnetic resonance imaging scans (visceral or lymph node disease). Lymph nodes in the pelvis must measure at least 1.5 centimeter in a short axis to be considered target lesion according to the modified Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 based on the Prostate Cancer Working Group 2 (PCWG2) criteria
* Castration-resistant prostate cancer (PC) demonstrated during continuous androgen deprivation therapy (ADT), defined as 3 rises of prostate-specific antigen (PSA), at least 1 week apart, with the last PSA greater than or equal to (>=) 2 nanogram per milliliter (ng/mL)
* Prior hormonal interventions (including 1st generation antiandrogens [flutamide, bicalutamide, nilutamide], steroids, estrogens, finasteride, dutasteride) for PC are allowed. These therapies, except for gonadotropin releasing hormone analogs (GnRH) analogs and prednisone/prednisolone, must have been discontinued for minimally 4 weeks (2 weeks only for flutamide, nilutamide, or finasteride) before first dose of study drug

Exclusion Criteria:

* Known brain metastases
* Chemotherapy, or immunotherapy within 2 weeks or 5 half-lives of the drug prior to the first dose of study drug, whichever is longer, with a maximum of 4 weeks.
* Prior treatment with second-generation anti-androgens (example [eg], enzalutamide)
* Administration of an investigational therapeutic within 2 weeks or 5 half-lives of the drug prior to the first dose of study drug, whichever is longer, with a maximum of 4 weeks. And participant use radiopharmaceutical agents (eg, strontium-89) or investigational immunotherapy (eg, sipuleucel-T) within 12 weeks prior to the first dose of study drug
* Prior treatment with cytochrome 17 inhibitors (eg, abiraterone acetate, orteronel, galeterone, systemic ketoconazole)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 19 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Plasma Concentration of Apalutamide | Predose; postdose up to 168 hours (hrs) (Cycle1 Day 7), Cycle 2 (pre-dose; on Day 1 and 15 of cycle 2) and Cycle 3 (pre-dose; up to 24 hrs post-dose). Each cycle is of 28 days
  Plasma concentration of apalutamide will be reported.
Number of Participants with Adverse Events | Up to 30 days of last study treatment (approximately 18 months)
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

SECONDARY OUTCOMES:
Change from Baseline in Serum Prostate Specific Antigen (PSA) at Weeks 4 and 12 | Baseline, at Weeks 4 and 12 or earlier for those who discontinue therapy (up to approximately 4 months).
  Change from baseline in serum PSA levels will be determined.
Maximal Decline in Prostate Specific Antigen | Up to 30 days of last study treatment (approximately 18 months)
  Maximal decline in PSA levels will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (4):
- China (4):
  - Peking University Third Hospital, Beijing
  - Beijing Cancer Hospital of Peking University, Beijing
  - Jiangsu Cancer Hospital, Nanjing
  - Fudan Cancer Hospital, Shanghai